CLINICAL TRIAL: NCT05571579
Title: Biological Collection of Brain Tumors - GLIOLI Collection
Brief Title: Biological Collection of Brain Tumors
Acronym: GLIOLI
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0813
Record Dates: First submitted 2022-10-03; First posted 2022-10-07 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Brain Tumor
Keywords: Brain tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * 1 tube of blood of 4 mL on dry tube with or without gel,
  * 2 tubes of blood of 4 mL on EDTA tube, If CSF collected for diagnosis is available, it can be sent for storage in the collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- brain tumors
  Interventions: Biological: blood and/or csf collection

INTERVENTIONS:
Biological: blood and/or csf collection — blood and/or collection
  Only once :
  * 1 tube of blood of 4 mL on dry tube with or without gel,
  * 2 tubes of blood of 4 mL on EDTA tube, If CSF collected for diagnosis is available, it can be sent for storage in the collection.

SUMMARY:
The objective of this study is to build a collection of biological samples from patients with brain tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose diagnosis of brain tumor has been confirmed.
* Adult patients, from 18 years old and without upper age limit
* Patient affiliated to a social security scheme or equivalent.
* Patient able to consent, having dated and signed an informed consent

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patient under guardianship or curators.
* Persons deprived of their liberty by a judicial or administrative decision

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with brain tumor
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2033-11-22 (Estimated); Study Completion 2033-11-22 (Estimated)

PRIMARY OUTCOMES:
number of biological samples | 10 years
  number of biological samples

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Bron, Rhône, France

IPD SHARING:
Plan to Share IPD: No